CLINICAL TRIAL: NCT04519580
Title: Improved Diagnostics and Monitoring of Polymyalgia Rheumatica
Status: Active, not recruiting | Type: Observational
Sponsor: Kresten Krarup Keller (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kresten Krarup Keller, MD, PhD, Central Jutland Regional Hospital
Organization: Central Jutland Regional Hospital (Other)
Other Study IDs: IMPROVE PMR
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Polymyalgia Rheumatica; Giant Cell Arteritis; Adrenal Insufficiency
Keywords: Positron emission computed tomography; Ultrasound
MeSH Terms: conditions — Polymyalgia Rheumatica; Giant Cell Arteritis; Adrenal Insufficiency | interventions — Positron Emission Tomography Computed Tomography; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected polymyalgia rheumatica: The study investigates patients with suspected polymyalgia rheumatica (PMR). For Patients where the PMR diagnosis is dismissed, the study terminates after the first visit. Patients diagnosed with PMR will be treated with prednisolone with taper corresponding to usual care. At baseline all patients will have medical history taken, physical examination, blood drawn, Synacthen® test, PET/CT, and ultrasound performed. Physical examination, PET/CT, and ultrasound are repeated after 8 weeks of prednisolone treatment while the patients iare on 10 mg prednisolone as well as after prednisolone taper two weeks later, where Synachten® test is also performed. After 10 weeks prednisolone is restarted at 10 mg and the patient is followed by their general practitioner or at the department of rheumatology, where prednisolone is tapered according to usual care. Patients are invited to a follow up visit after one year.
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — FDG-PET/CT at baseline, week 8 and week 10.
  Other Names: Ultrasound

SUMMARY:
Background: Polymyalgia rheumatica (PMR) is characterised by pain of the proximal muscles, general symptoms, and raised inflammatory markers. Treatment with prednisolone has several adverse effects. PMR is an exclusion diagnosis, and methods to diagnose and monitor the disease are lacking.

Objective: To investigate if ultrasound and PET/CT can be used to diagnose and monitor PMR. In addition, the importance of prednisolone induced adrenal insufficiency is investigated.

Methods: It is a prospective observational study in patients suspected of PMR. Patients diagnosed with PMR continue in the study. Ultrasound and PET/CT are performed at baseline, after 8 weeks on prednisolone, and after 10 weeks during a short prednisolone break. Adrenal insufficiency is investigated five times throughout the study. After one year the PMR diagnosis is confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of PMR.
* Age above 50
* Pain of the proximal muscles.

Exclusion Criteria:

* Peroral, intraarticular, intramuscular and dermal application of glucocorticoids within the last 3 month.
* Previous prednisolone treatment for GCA/PMR
* Unable to give consent.
* Symptoms of GCA (headache, jaw claudication, vision disturbances).
* Active malignant cancers within the last 5 years (except basal cell carcinoma).
* Other inflammatory rheumatic diseases (eg. rheumatoid arthritis, polymyositis, spondyloarthritis, psoriatic arthritits, gout).
* Uncontrolled diseases (eg severe active astma, cardiac disease with NYHA class IV)
* Treatment with peroral oestrogens, aminogluthethimid, trilostan, ketoconazole, fluconazol, etomidate, phenobarbital, phenytoin, rifampicin, metyrapon, mitotane.
* Known primary or secondary adrenal insufficiency.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients suspected for PMR.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PMR diagnosis at baseline with PET/CT | Baseline
  Sensitivity and specificity of PET/CT for PMR diagnosis at baseline with the clinical diagnosis after 1 year as reference standard and patients not diagnosed with PMR serving as controls.

SECONDARY OUTCOMES:
PMR diagnosis at week 8 with PET/CT | 8 weeks
  Sensitivity and specificity of PET/CT for PMR diagnosis at week 8 with the clinical diagnosis after 1 year as reference standard and patients not diagnosed with PMR serving as controls.
PMR diagnosis at week 10 with PET/CT | 10 weeks
  Sensitivity and specificity of PET/CT for PMR diagnosis after one week of discontinuation of glucocorticoids (week 10) with the clinical diagnosis after 1 year as reference standard and patients not diagnosed with PMR serving as controls.
Change in Ultrasound parameters from baseline to week 8 | 8 weeks
  Change in presence and thickness of subdeltoid bursitis and biceps tenosynovitis from baseline to week 8.
Change in Ultrasound parameters from week 8 to week 10 | 10 weeks
  Change in presence and thickness of subdeltoid bursitis and biceps tenosynovitis from week 8 to week 10.
Change in PET/CT parameters from baseline to week | 8 weeks
  Change in PET/CT parameters from baseline to week 8.
Change in PET/CT parameters from week 8 to week 10. | 10 weeks
  Change in PET/CT parameters from week 8 to week 10.
Frequency of adrenal insufficiency at week 10. | 10 weeks
  Frequency of adrenal insufficiency at week 10.
Presence of adrenal insufficiency at week 10 as a predictor of prednisolone cessation at one year. | 12 months
  Presence of adrenal insufficiency at week 10 as a predictor of prednisolone cessation at one year.
Presence of adrenal insufficiency at week 10 as a predictor of relapse at week 10. | 10 weeks
  Presence of adrenal insufficiency at week 10 as a predictor of relapse at week 10.
Frequency of adrenal insufficiency | 18 months
  Frequency of adrenal insufficiency after 1 and 1.5 years.
Lean boyd weight | 18 months
  Lean body weight adjusted prednisolone dose as a predictor of adrenal insufficiency.
Hypercortisolism as predictor of adrenal insufficiency. | 18 months
  Clinical and biochemical signs of hypercortisolism as predictor of adrenal insufficiency.
Change in clinical parameters week 8. | 8 weeks
  Change in clinical parameters from baseline to week 8.
Change in clinical parameters week 10. | 10 weeks
  Change in clinical parameters from week 8 to week 10.
Frequency of GCA | 12 months
  Frequency of GCA at diagnosis and during follow up
Change in PROM's from baseline to week 8. | 8 weeks
  Change in PROM's from baseline to week 8.
Change in PROM's from week 8 to week 10. | 10 weeks
  Change in PROM's from week 8 to week 10.
Change in PROM's from baseline to 1 year. | 12 months
  Change in PROM's from baseline to 1 year.
Sensitivity and specificity of CRP for PMR diagnosis at week 10. | 10 weeks
  Sensitivity and specificity of CRP for PMR diagnosis at week 10.
Level of inflammatory markers in PMR patients at baseline vs. week 8. | 8 weeks
  Level of inflammatory markers in PMR patients at baseline vs. week 8.
Level of inflammatory markers in PMR patients vs. non PMR patients at baseline. | Baseline
  Level of inflammatory markers in PMR patients vs. non PMR patients at baseline.
Change in expression levels of clock gene mRNA as marker of prednisolone-induced changes in sleep, lipid levels and glycated hemoglobin. | 1 year
  Change in expression levels of clock gene mRNA as marker of prednisolone-induced changes in sleep, lipid levels and glycated hemoglobin.
Percentage of patients with concomitant GCA and PMR after 3 and 5 years. | 5 Years
  Percentage of patients with concomitant GCA and PMR after 3 and 5 years.
Percentage of patients receiving prednisolone after 3 and 5 years. | 5 Years
  Percentage of patients receiving prednisolone after 3 and 5 years.
PET/CT measures at baseline as a predictor of prednisolone treatment after 3 and 5 years. | 5 Years
  PET/CT measures at baseline is measured with Standard Uptake Value and dichrotone evaluation for PMR (PMR +/-)
Changes in PET/CT parameters from baseline to week 8 as predictor of prednisolone treatment after 3 and 5 years | 5 Years
  PET/CT changes from baseline to 8 weeks in Standard Uptake Value and dichrotone evaluation for PMR (PMR +/-) will be evaluated.
Adrenal insufficiency as a predictor of prednisolone treatment after 3 and 5 years. | 5 Years
  Adrenal insufficiency (+/-) will be evaluated with synachten test 4-5 times during the first 1,5 year of the study. At least one positive value will contribute to the parameter.
Changes in US findings from baseline to week 8 as predictor of prednisolone treatment after 3 and 5 years | 5 Years
  Ultrasound dichrotone changes from baseline to week 8 will be evaluated (positive/negative for bursitis/artritis)

CONTACTS AND LOCATIONS:
Overall Officials: Kresten Keller, MD, Principal Investigator — Department of Rheumatology, Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Department of Rheumatology, Aarhus University Hospital, Aarhus
  - Department of Rheumatology, Horsens Regional Hospital, Horsens
  - Diagnostic Centre, Silkeborg Regional Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaster T, Nielsen AW, Hansen SB, Donskov AO, Nielsen MK, Hansen IT, Nielsen BD, Kjaer SG, Blegvad-Nissen J, Moller Sorensen C, Hauge EM, Jorgensen JOL, Keller KK. Repeated short corticotropin testing in patients with polymyalgia rheumatica. Rheumatology (Oxford). 2025 Nov 20:keaf614. doi: 10.1093/rheumatology/keaf614. Online ahead of print. PMID 41264768
- [Derived] Nielsen AW, van Praagh GD, van der Geest KSM, Hansen IT, Nielsen BD, Kjaer SG, Blegvad-Nissen J, Rewers K, Sorensen CM, Brouwer E, Hauge EM, Gormsen LC, Slart RHJA, Keller KK. Whole-body and site specific [18F]FDG uptake patterns on PET/CT have limited value in differentiating between polymyalgia rheumatica and other inflammatory diseases: two cohorts of treatment-naive suspected polymyalgia rheumatica. EJNMMI Res. 2025 Apr 30;15(1):51. doi: 10.1186/s13550-025-01233-7. PMID 40307615
- [Derived] Nielsen AW, Hauge EM, Hansen IT, Nielsen BD, Kjaer SG, Blegvad J, Rewers K, Moller Sorensen C, Gormsen LC, Keller KK. Low incidence of late-onset giant cell arteritis during the first year in patients with polymyalgia rheumatica-a repeated imaging study. Rheumatology (Oxford). 2025 Apr 1;64(4):2193-2198. doi: 10.1093/rheumatology/keae463. PMID 39180419
- [Derived] Nielsen AW, Hansen IT, Nielsen BD, Kjaer SG, Blegvad-Nissen J, Rewers K, Sorensen CM, Hauge EM, Gormsen LC, Keller KK. The effect of prednisolone and a short-term prednisolone discontinuation for the diagnostic accuracy of FDG-PET/CT in polymyalgia rheumatica-a prospective study of 101 patients. Eur J Nucl Med Mol Imaging. 2024 Jul;51(9):2614-2624. doi: 10.1007/s00259-024-06697-8. Epub 2024 Apr 2. PMID 38563881